CLINICAL TRIAL: NCT00006812
Title: Phase II Evaluation Of Capecitabine In Recurrent Platinum-Sensitive Ovarian Or Primary Peritoneal Cancer
Brief Title: Capecitabine in Treating Patients With Recurrent Ovarian Epithelial or Primary Peritoneal Cavity Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000068330; GOG-0146L
Record Dates: First submitted 2000-12-06; First posted 2004-03-17 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2005-11

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Capecitabine

INTERVENTIONS:
Drug: capecitabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of capecitabine in treating patients who have recurrent ovarian epithelial or primary peritoneal cavity cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of capecitabine in patients with recurrent, platinum-sensitive ovarian epithelial or primary peritoneal cavity cancer.
* Determine the nature and degree of toxicity of this drug in this patient population.

OUTLINE: This is a multicenter study.

Patients receive oral capecitabine twice daily for 14 days. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 22-60 patients will be accrued for this study within 6-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven recurrent ovarian epithelial or primary peritoneal cavity cancer
* Measurable disease

  * At least 1 unidimensionally measurable lesion
  * Ascites and pleural effusions are not considered measurable disease
* Prior therapy must include 1 platinum-based chemotherapy regimen for primary disease containing carboplatin, cisplatin, or another organoplatinum compound

  * Treatment-free interval of 6-12 months after response to platinum therapy
* Not eligible for higher priority GOG protocol

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* GOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least lower limit of normal

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine clearance at least 50 mL/min

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No neuropathy (sensory and motor) greater than grade 1
* No other malignancy within the past 5 years except nonmelanoma skin cancer
* No concurrent active infection requiring antibiotics

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior biologic or immunologic therapy
* No concurrent prophylactic filgrastim (G-CSF)

Chemotherapy:

* See Disease Characteristics
* If no prior therapy with paclitaxel, a second regimen including paclitaxel allowed
* No prior capecitabine or fluorouracil
* No prior chemotherapy for recurrent or persistent disease, including pretreatment with initial chemotherapy regimens
* Recovered from prior chemotherapy

Endocrine therapy:

* At least 1 week since prior hormonal therapy directed at malignant tumor
* Concurrent continuation of hormone replacement therapy allowed

Radiotherapy:

* At least 3 weeks since prior radiotherapy and recovered
* No prior radiotherapy to site(s) of measurable disease
* No prior radiotherapy to more than 25% of bone marrow

Surgery:

* Recovered from prior surgery

Other:

* No prior cancer treatment that would preclude study therapy
* No concurrent amifostine or other protective reagents

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-03; Primary Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agustin Garcia, MD, Study Chair — University of Southern California
Locations (31):
- United States (30):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of Colorado Cancer Center, Denver, Colorado
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Radiation Oncology Branch, Bethesda, Maryland
  - Tufts University School of Medicine, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
- Tom Baker Cancer Center - Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Result] Garcia AA, Blessing JA, Lenz HJ, Darcy KM, Mannel RS, Miller DS, Husseinzadeh N; Gynecologic Oncology Group. Phase II clinical trial of capecitabine in ovarian carcinoma recurrent 6-12 months after completion of primary chemotherapy, with exploratory TS, DPD, and TP correlates: a Gynecologic Oncology Group study. Gynecol Oncol. 2005 Mar;96(3):810-7. doi: 10.1016/j.ygyno.2004.11.037. PMID 15721430